CLINICAL TRIAL: NCT00714259
Title: UAB 0775 Phase II Trial of Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation Protocol From HLA Matched Related Donors for The Treatment of Patients With Low Grade B Cell Malignancies
Brief Title: Non-Myeloablative Allogeneic HSCT From HLA Matched Related or Unrelated Donors for the Treatment of Low Grade B Cell Malignancies
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Accrual goals could not be met within a timely manner
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Racquel Innis-Shelton, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F080429003; UAB-0775 (Other: UAB Cancer Center study number)
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma; CLL / SLL; Non Hodgkin's Lymphoma; Waldenstroms; Mantle Cell Lymphoma
Keywords: Low Grade B Cell Malignancies; nonmyeloablative transplant; allogeneic
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Leukemia, B-Cell | interventions — fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non Myeloablative Treatment (Other): Non-myeloablative Transplant Conditioning Chemotherapy :
  Fludarabine - 30 mg/m2/day x 3 days Total Body Irradiation - 200cGy x1 dose Infusion of Stem Cells - On Day 0 pts will received an infusion of HLA matched sibling donor stem cells. Dose is determined by the volume of cells obtained from donor. Minimum dose is 2x10*6 CD34+ cells per kilogram of recipient weight.
  Interventions: Drug: Fludarabine; Radiation: Total Body Irradiation; Other: Infusion of Stem Cells

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2/day x 3 days
Radiation: Total Body Irradiation — TBI 200cGy x1 dose on transplant day
Other: Infusion of Stem Cells — On Day 0 pts will received an infusion of HLA matched sibling donor stem cells. Dose is determined by the volume of cells obtained from donor. Minimum dose is 2x10*6 CD34+ cells per kilogram of recipient weight.

SUMMARY:
A non-myeloablative treatment strategy and uniform selection criteria will enable patients with a variety of low grade B-Cell malignancies to attain long term disease control without unacceptably high treatment related mortality.

DETAILED DESCRIPTION:
Non myeloablative transplant aims to achieve the immunological advantage of graft versus tumor effect as conventional myeloablative therapy without causing high treatment related toxicities. Non myeloablative transplant has been gaining wider acceptance as a way to achieve longer disease free and over all survival in patients with low grade B-cell malignancies, which otherwise is an incurable disease. Recent studies of non-myeloablative HSCT have demonstrated the powerful effect of graft versus leukemia alone against myeloma and other malignant B-cell malignancies if the transplant is performed for low grade, low volume disease.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III non-progressive disease Multiple Myeloma.
* CLL/SLL, and low grade Hodgkin Lymphomas that are in a very good partial response or complete response with non-progressive disease.
* ≤ 70 years old.
* Eligible and willing HLA matched related donor.
* Bilirubin <2xULN.
* ALT and AST <3xULN.
* LVEF > 40%.
* Creatinine Clearance >40mL/min.
* Pulmonary function DLCO corrected to ≥ 70%.
* Minimum performance score of 70%.
* Platelet count >130 x103 micro L.
* LDH ≤1.5xULN.
* No proceeding co-morbid condition that significantly increases the risk of severe regimen related toxicity.
* No uncontrolled infections.

Exclusion Criteria:

* Age >70 years old.
* Performance status <70%.
* Uncontrolled infections or is HIV positive
* Prior malignancies that are felt to have a <80% probability of being cured.
* Pregnant, breastfeeding, or refuse to use contraceptive techniques during and for 12 months following transplant.
* Prior Allograft
* History of rapidly growing disease at diagnosis or at any progression or have MDS.
* No eligible and willing HLA matched donor.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P. Vaughan, MD, Principal Investigator — University of Alabama in Birmingham
Locations (1):
- University of Alabama in Birmingham BMT/CT Program Outpatient Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Trial: Single Arm Intervention trial as noted in interventions section
  Fludarabine: Fludarabine 30 mg/m2/day x 3 days
  Total Body Irradiation: TBI 200cGy x1 dose on transplant day
  Infusion of Stem Cells: On Day 0 pts will received an infusion of HLA matched sibling donor stem cells. Dose is determined by the volume of cells obtained from donor. Minimum dose is 2x10*6 CD34+ cells per kilogram of recipient weight.
Period: Overall Study
Arm/Group | Single Arm Trial
Started | 5
Completed | 3
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Progressive Free Survival Post Transplant
Description: subjects surviving without disease progression at 100 days after transplant as evidenced by decreased disease and no new disease showing on radiologic scans and / or bone marrow pathology.
Time Frame: 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 5
participants | 4

2. Secondary Outcome: Non-relapse Treatment Related Mortality
Description: Death related to treatment without relapse within 100 days after transplant
Time Frame: Within 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 5
participants | 0

3. Secondary Outcome: Number of Participants With Detectable Donor Chimerism at up to 100 Days Post Transplant
Description: Measured by number of participants that have chimerism study results that show the number of donor cells and the number of recipient cells present in the blood after post-transplant lymphocyte infusions continue to be predominately either donor or recipient.
Time Frame: Post transplant up to 100 days post transplant
Measure: Number; unit: participant
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 5
participant | 1

4. Secondary Outcome: Composite Incidence of Acute and Chronic Graft Versus Host Disease
Time Frame: Up to 100 days post transplant.
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 5
participants | 2

5. Primary Outcome: Progressive Free Survival Post Transplant
Description: Subjects surviving without disease progression 180 days after transplant as evidenced by decreased disease and no new disease showing on radiologic scans and / or bone marrow pathology.
Time Frame: 180 days post transplant
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 4
participants | 4

6. Primary Outcome: Progressive Free Survival Post Transplant
Description: Subjects surviving without disease progression 365 days after transplant as evidenced by decreased disease and no new disease showing on radiologic scans and / or bone marrow pathology.
Time Frame: 365 days post transplant
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 4
participants | 4

7. Primary Outcome: Progression Free Survival Post Transplant
Description: Subjects surviving without disease progression 2 years after transplant as evidenced by no new disease showing on radiologic scans and / or bone marrow pathology.
Time Frame: 2 years post transplant
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 4
participants | 2

ADVERSE EVENTS:
Arm/Group | Single Arm Trial
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Trial (N=5)
RSV pneumonia Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Klebsiella pneumonia Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia not otherwise specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No